CLINICAL TRIAL: NCT01352949
Title: Stereophotogrammetry of the Torso in Healthy Individuals and Patients With Scoliosis, Chest Wall Deformations, or Obesity
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 110120; 11-CC-0120
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-05-09

CONDITIONS: Bone Diseases; Obesity; Healthy Volunteers
Keywords: Anthropometry; Stereophotogrammetry; Torso; Natural History
MeSH Terms: conditions — Bone Diseases; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Healthy volunteers without scoliosis or obesity
- Obesity: Healthy volunteers with obesity
- Scoliosis: Healthy volunteers with scoliosis but no obesity

SUMMARY:
Background:

- Stereophotogrammetry (SP) uses four sets of digital cameras to generate a three-dimensional computer image. Unlike other types of evaluations which require radiation, SP only uses computer images to learn more about physical deformities such as scoliosis or about the placement of fat on the body. To refine the SP process, researchers are interested in collecting images and body data from individuals with skeletal structural problems such as scoliosis or chest wall deformities, individuals who are overweight or obese, and healthy volunteers.

Objectives:

- To use stereophotogrammetry to study different individual body types and refine existing imaging techniques.

Eligibility:

- Individuals at least 2 years of age who have spine, rib, or chest wall deformities; are overweight or obese (body mass index greater than 25); or are healthy volunteers.

Design:

* Participants will be screened with a physical examination and medical history. The physical examination will include measurements of range of motion and joint mobility, torso width and length, and other observational data.
* Healthy volunteers and participants in the obesity group will also have bioelectric spectroscopy (bioimpedance), which uses an additional machine to measure how fat is spread in different parts of the body.
* After the physical examination has been completed, participants will have SP photographs taken. Participants will be asked to remove all clothing from the torso, stand with arms raised at the center of four cameras, and remain still while several images are taken. A complete image takes less than 1 second.
* Participants with spine or rib deformities, or who are in the obesity group, may also volunteer to return for followup SP imaging, once a year for 5 years, to study progress over time.

DETAILED DESCRIPTION:
Objective

The primary objective of this project is to determine which outcome measures derived from analysis of SP images are reliable within the healthy population and can distinguish between healthy volunteers and those with scoliosis, chest wall deformities, and obesity. Secondary objectives include comparing SP outcome measures with clinical and radiographic measures to test concurrent validity and to determine if the SP outcome measures correlate with clinical and radiographic measures taken over time. The ultimate goal is to develop SP as a measurement tool to be employed in clinical research involving the study of scoliosis, rib and chest deformities and the truncal distribution of adiposity.

Study population

The population for this study consists of healthy volunteers, persons with scoliosis and/or chest wall deformities, and persons with obesity. Men and women of all races, ethnicities, and ages greater than two years may participate.

Design

This project will be carried out in three phases. In Phase I, we will analyze images of healthy volunteers captured by the SP scoliosis and chest-wall deformity ( scoliosis ) software to identify the outcome measures that show minimal or no variance. We will also examine if healthy volunteers gender, age, height, and BMI contribute to the differences of these outcome measures.

In Phase IIa, images captured from subjects with scoliosis and/or chest wall deformities will be processed by scoliosis software to determine the set of meaningful variables (those that show significant differences between the two populations). In Phase IIb, images captured of healthy volunteers will be processed using obesity software to determine the set of variables showing minimal or no variance among the data from healthy volunteers when controlling for the effects of potential confounders. Variables that continue to have minimal or no variance will be considered meaningful with respect to obesity analysis software. Those variables achieved from obesity image analysis will be compared to the set from the healthy volunteers to determine which variables show significant differences between the healthy volunteer and obese subjects.

In Phase III, healthy participants, scoliosis/chest wall deformity, and obesity participants who are scheduled to return to NIH as part of another NIH protocol will be invited to return for yearly re-imaging up to a total of five years in order to analyze changes over time and compare them with concurrent radiographic measures.

Outcome measures

The purpose of the study is to develop outcome measures for use in future research. These outcome measures will be developed from software which analyzes images derived from the stereophotogrammetry system.

ELIGIBILITY:
* INCLUSION CRITERIA:

  * All subjects greater than 2 years of age, genders, and ethnicities will be eligible so long as they can cooperate with physical examination and imaging procedures.
  * Subjects must be able to stand independently for imaging. This limits enrollment to subjects 2 years of age and older.
  * Subjects must agree to capture of image of their bare torso above the waist
  * Healthy volunteers must be without scoliosis, or chest wall deformities, and with BMI below overweight range. For adults, BMI must be less than or equal to 25. BMI for children and adolescents will be corrected according to the guidelines designated by the Centers for Disease Control and Prevention found in Appendices 2 (boys) and 3 (girls).
  * Adults with BMI less than or equal to 25 and children and adolescents with adjust BMI below the overweight range AND with imaging confirmed scoliosis and/or chest wall deformities will be recruited from participants in NIH intramural protocols or referred by outside physicians and will be eligible to participate in phase IIa of the study.

    * Adults (subjects who are 18 years of age or older), must either present a previously obtained clinical standing scoliosis xray film dated no more than 12 months prior to the study visit or obtain a scoliosis series x-ray at the National Institutes of Health Clinical Center to provide confirmation of scoliosis. Therefore, xrays may be done for research purposes in adults if there is prior imaging indication but no scoliosis series xray films taken within the last 12 months.
    * Children must present a previously obtained clinical standing scoliosis film dated no more than six months prior to the study visit to provide radiological confirmation of scoliosis. No xrays will be done for research purposes.
    * Volunteers who have undergone spinal fusion surgery must show a postoperative film that shows that the instrumentation is intact and that desired spinal fusion has occurred. Xrays may be done for research purposes in adults if there is prior imaging indication but no scoliosis x-ray series films taken within the last 12 months.
  * Subjects with BMI greater than 25 (or for children and adolescents defined according to Centers for Disease Control and Prevention guidelines as "overweight") AND without deformities of the torso will be eligible to participate in phase IIb, the obesity portion of the study.
  * Subjects with deformities of the torso OR with BMI greater than 25 may be eligible to participate in Phase IIIa or IIIb and be followed yearly over the course of five years

    * Subjects with scoliosis and/or chest wall deformities that are followed over the course of the five years must provide clinically obtained films with at least a difference of a year between the current and previous films. In adults, if the curve changes, it is clinically indicated to get a follow-up film and subsequent scoliosis xray films may be taken at the NIH CC. Those who do not require clinical films cannot be included in the scoliosis/chest wall deformities group followed over time.
    * For subjects of BMI greater than 25, volunteers will be invited to be followed over time using SP if they have a change in their body composition over time (if they have not yet attained physical maturity, if they participate in weight loss program, or report a significant weight gain).

EXCLUSION CRITERIA:

* Subjects unable to tolerate having points on the torso marked with a surgical ink marker
* Subjects with contact or respiratory isolation status
* Subjects with pacemakers or other electrical or conducting metal medical devices implanted in their torso will not be able to participate in the normal volunteer and obesity groups due to contraindication to participation in bioelectric spectroscopy testing.
* Subjects with electrical or conducting metal medical devices in their arms or legs that are not limited to one side of the body will not be able to participate in the normal volunteer and obesity groups because it will cause data distortion in the bioelectric spectroscopy testing.
* Subjects who are unable to tolerate stroboscopic camera flash
* Subjects who are employees/staff of the NIH Clinical Center Rehabilitation Medicine Department.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population for this study consists of healthy volunteers, persons with scoliosis and/or chest wall deformities, and persons with obesity. Men and women of all races, ethnicities, and ages greater than two years may participate.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2011-06-02 (Actual)

PRIMARY OUTCOMES:
Output variables provided by the Matlab stereophotogrammetry analysis program | after accrual of 50 subjects, 100 subjects, and all subjects
  Measures derived from mathematical analysis of cross sections of the 3d torso computer model
Other variables calculated from the Matlab stereophotogrammetry output variables | after accrual of 50 subjects, 100 subjects, and all subjects
  Variables calculated by comparing and connecting the outputs of individual cross sectional analyses described above.

SECONDARY OUTCOMES:
pelvic obliquity | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for scoliosis/chest-wall deformities
AP chest diameter | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for scoliosis/chest-wall deformities
Adam s forward bending test | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for scoliosis/chest-wall deformities
rib symmetry | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for scoliosis/chest-wall deformities
finger-floor test | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for obesity
Schober test | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for obesity
stand and reach | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for obesity
WHR | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for obesity
leg length discrepancies | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for scoliosis/chest-wall deformities
pectus carinatum | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for scoliosis/chest-wall deformities
chest circumference | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for scoliosis/chest-wall deformities
pectus excavatum | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for scoliosis/chest-wall deformities
BMI | after accrual of 50 subjects, 100 subjects, and all subjects
  physical parameters which will be measured in order to perform tests of concurrent validity for obesity

CONTACTS AND LOCATIONS:
Overall Officials: Galen O Joe, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-CC-0120.html